CLINICAL TRIAL: NCT06250491
Title: Effects of Deep rTMS in Neuropathic Pain or Fibromyalgia : a Bicenter Randomized Sham Controlled Study
Brief Title: Deep rTMS (H-coil) for Neuropathic Pain or Fibromyalgia
Acronym: H-FINEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nadine ATTAL (Other)
Responsible Party: Sponsor-Investigator, Nadine ATTAL, Clinical Professor, Hospital Ambroise Paré Paris
Organization: Hospital Ambroise Paré Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-A00902-43
Record Dates: First submitted 2024-01-23; First posted 2024-02-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Neuropathic Pain; Fibromyalgia
MeSH Terms: conditions — Neuralgia; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS (Experimental): Deep rTMS with H coil targeting the motor cortex bilaterally
  Interventions: Device: Deep active rTMS with Hesed coil; Device: Sham rTMS with Hesed coil
- Sham rTMS (Placebo Comparator): Sham rTMS with H coil targeting the motor cortex bilaterally
  Interventions: Device: Deep active rTMS with Hesed coil; Device: Sham rTMS with Hesed coil

INTERVENTIONS:
Device: Deep active rTMS with Hesed coil — This brain neurostimulation method targets the motor cortex bilaterally
Device: Sham rTMS with Hesed coil — This brain sham neurostimulation method targets the motor cortex bilaterally

SUMMARY:
This study will investigate the efficacy and safety of "deep" rTMS on neuropathic pain or fibromyalgia. It will be randomized and sham controlled and will last 3 months. Patients will be randomized to receive acctive rTMS or sham rTMS and will receive repeated rTMS sessions (5 daily sessions then one session per week then every 2 to 3 weeks for up to 10 weeks).

DETAILED DESCRIPTION:
This double blind sham controlled parallel group bicenter study will assess the efficacy and safety of repeated sessions of deep rTMS using H coil in patients with neuropathic pain or fibromyalgia. Primary outcome will be % of pain relief at week 13.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain ≥ 6 months, at least 4/10 on a 0-10 NRS, present every day or nearly every day
* Neuropathic pain (confirmed with Douleur Neuropathique en 4 questions and international criteria from NeuPSIG) or fibromyalgia (revised ACR criteria)
* Stable concomitant medications for pain for at least one month
* Able to fill out questionnaires and understand and speak French

Exclusion Criteria:

* Contraindications to rTMS
* Prior treatment with rTMS
* Progressive severe condition (eg cancer)
* Psychosis
* Psychoactive drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Effects of rTMS versus sham rTMS on pain relief at 13 weeks | 13 weeks
  Pain relief scale from the Brief Pain Inventory rated from 0 to 100 %

SECONDARY OUTCOMES:
Effects of rTMS vs sham on average pain intensity | Each follow up visit at the pain center for up to 13 weeks
  Average pain intensity from the Brief Pain Inventory rated from 0 to 10 on a 0-10 numerical pain scale
Effects of rTMS vs sham on pain interference | Baseline then each follow up visit at the pain center for up to 13 weeks
  pain interference from Brief Pain Inventory rated from 0 to 70 (total score)
Effects of rTMS vs sham on quality of life | Baseline then each follow up vist at the pain center for up to 13 weeks
  Euroqol scale which includes 5 dimensions of quality of life and a 0-100 visual analog scale
Side effects of rTMS or sham | Each follow up visit at the pain center for up to 13 weeks
  Any side effects reported by the patients assessed at each visit after each treatment session and rated as mild, moderate or severe
Comparison of the efficacy of rTMS on the primary outcome between patients with neuropathic pain and fibromyalgia | Week 13
  Comparison of both populations on the pain relief scale from the Brief Pain Inventory (0-100 %)
Blinding assessment | 13 weeks
  Blindinq questionnaire at 13 weeks(end of the study)
Patient global impression of change | 13 weeks
  Patient global impression of change at 13 weeks (from much improved to much deteriorated)
Self-reported pain intensity | Baseline then every day at the same time of day (morning or evening)
  Average pain intensity from past 24 hours based on 0-10 numerical pain scale
Effects of rTMS versus sham on anxiety and depressive symptoms | Baseline then each follow up visit at the pain center for up to 13 weeks
  Anxiety and depressive symptoms of the Hospital Anxiety and Depressive scale rated from 0 to 21 for anxiety and 0 to 21 for depression
Effects of rTMS vs sham on pain as its worst from Brief Pain Inventory | Baseline then each follow up visit at the pain center for up to 13 weeks
  pain intensity on 0-10 numerical rating scale
Effects of rTMS vs sham on pain as its least from Brief Pain Inventory | Baseline then each follow up visit at the pain center for up to 13 weeks
  pain intensiy on 0-10 numerical rating scale
Effects of rTMS vs sham on sleep | Baseline then each follow up visit at the pain center for up to 13 weeks
  Sleep assessed using the sleep scale from the Medical Outcome Survey
Effects of rTMS vs sham on pain right now from Brief Pain Inventory | Baseline then each follow up visit at the pain center for up to 13 weeks
  pain intensiy on 0-10 numerical rating scale
Effects on Global Impression of change assessed by the clinician | 13 weeks (end of the treatment)
  Clinician global impression of change (from much improved to much deteriorated)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine ATTAL, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Inserm U987, Boulogne-Billancourt
  - Centre d'Evaluation et de Traitement de la douleur, Paris

IPD SHARING:
Plan to Share IPD: No